CLINICAL TRIAL: NCT04396314
Title: Effectiveness of Basic Body Awareness Therapy in Survivors of Covid-19, Health Workers and Women Suffering From Gender-based Violence Regarding Post-traumatic Stress Disorders: A Randomized Clinical Trial
Brief Title: Effectiveness of Basic Body Awareness Therapy in Post-traumatic Stress Disorders: A Randomized Clinical Trial
Acronym: BATEP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universitat de Lleida (Other)
Collaborators: Francesc Rubí Carnacea (Unknown)
Responsible Party: Principal Investigator, Cristina Bravo, PhD, Universitat de Lleida
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UL-002
Record Dates: First submitted 2020-05-15; First posted 2020-05-20 (Actual); Last update posted 2021-03-19 (Actual); Status verified 2021-03

CONDITIONS: PostTraumatic Stress Disorder
Keywords: Basic Body Awareness Therapy; physiotherapy; anxiety; depression
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Anxiety Disorders; Depression

STUDY DESIGN:
Intervention Model Description: randomized controlled clinical trial
Who Masked: Outcomes Assessor
Masking Description: The researcher will be blinded to group of participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Basic Body Awareness Therapy (Experimental): Basic Body Awareness Therapy (BBAT), a health oriented, multi-perspective and person-centred approach with a focus on the patient's resources, is a movement awareness training approach in physiotherapy, aiming to promote movement quality in daily life through self-exploration and self-experience enabling the learning of new movement habits. BBAT consists of a broad scope of movements in the following positions: lying, sitting, standing and walking. Relational movements are practiced in therapy with components such as rhythm, form, elasticity, flow, intention and voice
  Interventions: Behavioral: Basic Body Awareness Therapy
- Control (Active Comparator): The control group will be treatment for usual for PTSD. Pharmacological treatment is based in fluoxetine, paroxetine, sertraline and venlafaxine. Regarding non-pharmacological treatment the strongly recommendations are cognitive-behavioural therapy, cognitive processing therapy, cognitive therapy and prolonged exposure therapy
  Interventions: Behavioral: Psychological treatment

INTERVENTIONS:
Behavioral: Basic Body Awareness Therapy — Basic Body Awareness Therapy (BBAT), a health oriented, multi-perspective and person-centred approach with a focus on the patient's resources. It is a movement awareness training approach in physiotherapy, aiming to promote movement quality in daily life through self-exploration and self-experience enabling the learning of new movement habits
  Arms: Basic Body Awareness Therapy
Behavioral: Psychological treatment — Cognitive-behavioural therapy, cognitive processing therapy, cognitive therapy and prolonged exposure therapy
  Arms: Control

SUMMARY:
The aim of this randomized controlled clinical trial is to assess the effectiveness of Basic Body Awareness Therapy online in patients' survivors of Covid-19, health workers and women suffering from gender based violence regarding post-traumatic stress disorder in comparison with treatment as usual. The study will be multicentric in base Hospital Igualada and University of Lleida. The participants will be survivors of Covid-19 that had been inpatient in intensive care and health workers in first line with pandemia as doctors, nurse, physiotherapist, etc. More else, a new context emerge regarding gender based violence during the lockdown time. Outcomes variables will be measured regarding post-traumatic stress disorder, anxiety, depression, pain, quality of life and sleep. Fifty-four patients will be randomly assigned to a control group that will follow treatment as usual. The intervention group that will be received the same treatment adding Basic Body Awareness Therapy. The intervention will last 3 months twice a week at online format. At first month the intervention consisted of 12 movements and 15 min for sharing reflections about experiences. During the subsequent sessions, the treatment will be in group of 8 participants using the same methodology online. If the conditions of pandemia allow, the group will be presential in the health center at last month. Data analysis will performed using ANOVA of variables intragroup with repeated measurements. The analyses of the effects between groups will be performed throught ANOVA intergroup.

DETAILED DESCRIPTION:
This protocol of research is addressed to assess the effectiveness of Basic Body Awareness Therapy (BBAT) as physiotherapist intervention adjunct treatment as usual with the aim to improve the symptoms of post-traumatic stress disorder (PTSD) in survivors of Covid-19, health workers and women suffering from gender-based violence.

Nowadays the world lives a pandemic of unknown diseases with a high mortality and propagation. It results a huge number of patients admitted in intensive care unity. Health workers and patients suffering the fact of unknown the outcome of Covid-19 as such as, the treatment and prevention of it. The level of stress of that situation and the isolation could generate a breeding ground for develop the PTSD.

Post-traumatic stress disorder (PTSD) includes symptoms such as persistent re-experiencing, sleep pattern disorders, nightmares, hyperarousal, avoidance of stimuli associated with trauma or phobia occurring after a traumatic experience. Some situations that could provoke PTSD are sexual abuse, gender-based violence or danger of death situations such as wars, kidnapping.

Otherwise some diseases could trigger PTSD, in the epidermal necrolysis comprising Stevens-Johnson syndrome is usual the life-threatening reaction with a prevalence of 65% of patients presents PTSD and 29% possible clinical of PTSD. Also PTSD has been assessed in other situations such as gender-based violence in american students with a prevalence of 40.4%, moreover in war veterans the prevalence is between 11-20% while in war refugees the prevalence is 68% in Denmark. More else, a new context of gender-based violence emerges during the lockdown time in our society.

The pharmacological treatment for PTSD is based in fluoxetine, paroxetine, sertraline and venlafaxine. There is insufficient evidence to recommend for or against offering risperidone and topiramate. Regarding non-pharmacological treatment the strongly recommendations are cognitive-behavioural therapy, cognitive processing therapy, cognitive therapy and prolonged exposure therapy. Additionally, the clinical practice guideline conditionally recommends the use of brief eclectic psychotherapy, eye movement desensitization and reprocessing (EMDR), and narrative exposure therapy (NET) Basic Body Awareness Therapy (BBAT), a health oriented, multi-perspective and person-centred approach with a focus on the patient's resources, is a movement awareness training approach in physiotherapy, aiming to promote movement quality in daily life through self-exploration and self-experience enabling the learning of new movement habits. Understanding movement quality as the art of consciously being, doing and relating to oneself and others will result in more functional daily life, relationships and actions. The features of movement quality as a phenomenon in the physiotherapeutic context are classified into four perspectives- biomechanical, physiological, bio-psycho-social and existential. BBAT consists of a broad scope of movements in the following positions: lying, sitting, standing and walking. Relational movements are practiced in therapy with components such as rhythm, form, elasticity, flow, intention and voice. To gain more functional movement quality, the physiotherapist focuses the guidance on postural balance, free breathing, and awareness, seeking to integrate them into movement. This method is applied in conditions such as psychosomatic, eating disorders, schizophrenia, depression, chronic pain and PTSD.

Due to it is difficult to determinate the number of patients that will develop PTSD. Due to special circumstances of Spain without protective equipment, lack of health resources, changes in organization of health system and clinical guidelines and large etc. is predictable that health workers as nurses, doctors, physiotherapist and other professionals could develop PTSD, as well as, women suffering from gender violence. Studies about health workers shows that they are so susceptible to suffer PTSD in pandemic, crisis and emergency situations. It is predictable PTSD will appear as a high challenge in order to restore the health of survivors, health workers and women suffering from gender-based violence.

The aim of this study is to assess whether BBAT online adjunct with treatment as usual improves symptoms of PTSD in comparison of treatment as usual regarding level of anxiety, depression, quality of life, quality of sleep and pain.

Methods Hypothesis and general objectives: The project will be developed to answer questions about the effectiveness of BBAT regarding PTSD in survivors of Covid-19, health workers and women under gender violence. The hypothesis will be based on " the BBAT in survivors of Covid-19, health workers and women suffering violence as treatment adjunct of usual in comparison of treatment as usual alone, generate improvement of level of anxiety, depression, pain, quality of life and sleep diminishing the level of PTSD".

The general objectives will be assessed the response of survivors of Covid-10, health workers and women suffering violence to BBAT in comparison with treatment as usual. The specific objectives will be assessed the improvement of level of PTSD regarding anxiety, depression, quality of life and sleep and pain.

The study follows the Declaration of Helsinki and the "Guidelines for Good Clinical Practice". The clinical trial will be registered at ClinicalTrials.gov. According to the Helsinki Declaration, a specific informed consent will be used, which will be authorized by the local Ethical committee of Arnau de Vilanova Hospital and Igualada Hospital. Additionally, Royal Decree 3/2018 of 5th December which related to the data protection for the participants of the research, the data will be saved in an encrypted file. The ethical Committee of Clinical Research of Arnau de Vilanova of Lleida will approve the protocol. Clinical information, including clinical charts, pathology reports and working live will be available in anonymized data file that will be guarded by the main researcher.

Study participants According to the research protocol, the study will be conducted at a primary healthcare center. Participants will be eligible if 1) survivors of Covid-19, health workers and women suffering gender violence with level of post-traumatic stress disorder scale (DSM-V) moderate or severe, b) age >18 years, c) they could manage to stand in the position of "lying", "sitting", and "standing" without assistance. The exclusion criteria will be 1) they could not follow the intervention due to mental or physical health.

The sample size is determined according Argimon' formula of comparison of proportions. The psychological effectiveness as cognitive behaviour therapy is 60% of improvement of symptoms. The hypothesis will be arrived to 80% with a risk of 0.05 and statistical power of 95%. Due to data, the sample size will be of 23 participants by group. More else, the drop-out estimate is 15% and then, the group will be of 27 participants each one at least. The study is design multicentric and more than 27 participants are expected to be, the budget have the estimation of 81 participants in different settings.

A clinical trial will be conducted with two controlled and randomized parallel groups. The participants will have to be collected from the data base of mental health center of Igualada Hospital by a postdoc researcher and they will be invited to attend to an informational meeting. In this meeting, all patients willing to participate will have to sign a written informed consent form to participate in the trial and will have to full a socio-demographic questionnaire. The randomized process will complete using the software Epidat v 4.0. A number will assign to the participants, and then the program will generate two groups of numbers, the control and intervention groups. The results of randomizations will communicate by telephone to the participants. The study will start at September 2020 for 24 weeks, and all participants will assess at baseline, at 1 month of intervention, at end of the 3 months of treatment period and at 3 months follow-ups. Participants of both groups will be continued treatment as usual, which included pharmacological and psychological therapy. Participants in the control group will have the same exposure in time as the intervention group and will ask to maintain their lifestyle during the whole study and to refrain from starting any new regular physical activity. In case they could not maintain the same lifestyle during the study period, they will be asked to inform the researchers at any of the assessments.

Intervention: BBAT will be developed twice a week for 12 weeks online form. The intervention consisted in one month of individual treatment consisted on 12 movements. During the subsequent sessions, the participants joined in BBAT group sessions of 9 members each one. If the state of pandemic allows, the last 4 weeks the intervention will be on-site. The control group will follow the treatment as usual that consist in pharmacological treatment and cognitive based behaviour achieving by psychiatrist and psychologist.

Outcomes: the variables of study were in relation to PTSD, anxiety, and depression. The validate scales will be Davidson Trauma Scale (DTS) for PTSD, Visual Analogue Scale (VAS), Beck Depression Inventory (BDI) for depression, State Trait Anxiety Inventory (STAI) for anxiety, Short Form 36(SF-36) y Pittsburgh Scale (PS) for quality of life and sleep.

4.- Principal Investigator and team: The principal investigator will be Joan Blanco-Blanco, nurse specialist in geriatric and gerontology of Ministry of Education, Culture and Sports since 2014 and member of committee consultant of national group for studies and assessment of wound (GNEAUPP). Researcher of the Group of Studies on Society, Health, Education and Culture (GESEC) of the University of Lleida and collaborator of the Research Group on Health Cures (GRECS) of the Institute of Biomedical Research of Lleida (IRBLleida) in some projects with common interests. He is currently a professor at the Faculty of Nursing and Physiotherapy of the University of Lleida since 2009, where he received his PhD in 2013 (17/4/13) "cum laude", having directed 4 doctoral theses, more than 30 final papers and more than 15 final papers for his Master's degree. In this context, he has participated in several projects basically related to nursing practices in vulnerable groups, intergenerational learning through web platforms and problems related to aging, dependency and fragility, highlighting his work as a researcher in the European project ANIMATE and as a principal Researcher in the national project OTAGO. Reviewer of the journals: Clinical Nursing, Nutrients, Medicina Paliatiava, Journal of Advanced Nursing and Disability and Rehabilitation. In relation to team management, he was Dean of the Faculty of Nursing and Physiotherapy for 6 years, until 2019.

The following members also belong to the research team:

* Cristina Bravo Navarro has a research career in line with and favourable to this call, taking into account that she has already carried out a clinical trial with similar characteristics evaluating the effectiveness of BBAT in patients with fibromyalgia assessing variables related to pain, anxiety and depression. She has a doctorate in physiotherapy from the University of Lleida and a BBAT therapist from the University of Bergen (Norway). From her thesis "Effectiveness of Basal Body Awareness Therapy in patients suffering from fibromyalgia" from which numerous articles have been published in scientific journals.
* Dr. Joan Enric Torra-Bou is a post-doc researcher at the Faculty of Nursing and Physiotherapy of the University of Lleida with extensive experience in research who has directed a national project funded in 1998 file: 98/0483. He carried out his doctoral thesis on topics related to epidemiology. In 2017 he led a project funded by the Fundation Nursing and Society of the Barcelona College of Nursing PR-247/17. He also has numerous publications in the field of nursing and epidemiology.
* Dr. Daniel Catalán-Matamoros participates as an expert in BBAT, co-director of the International Master of Physiotherapy in BBAT at the University of Almería and has directed several doctoral theses on the effectiveness of BBAT in mental disorders and has numerous publications in the field of physiotherapy in mental health. He is also the president of the Spanish Association of Physiotherapists in Mental Health (www.fisioterapiasm.es) and has been a PI and researcher in projects funded by the European Commission and the National R&D Plan.
* Francesc Rubí-Carnacea participates as an expert in physical therapy in the field of chronic pain and therapeutic exercise. He has also participated in the development of several competitive projects and degree research works. He is a clinical physiotherapist with more than 25 years of experience in the psychosocial treatment of patients

  5.- Impact of the proposal: Regarding the scientific impact in relation within the challenge of health in pandemic circumstances it is necessary take care of health workers to cope the possible next pandemic situations and patients to be productive in society. The achievement of the objectives of the project will directly affect positively in the social economy of public health due the cost-effectiveness is significantly low in the physiotherapy intervention than pharmacology and psychology ones. Besides, the changes in lifestyle of patient probably will be long-lasting and it will suppose that patients will be autonomous, and they could manage their symptoms by oneself.

Also, if the hypothesis confirms there will be a new and safety treatment, even the researcher could hypothesize that movement awareness could effective to prevent the PTSD in next possible situations.

ELIGIBILITY:
Inclusion Criteria:

* a) survivors of COVID-19, health workers and women suffering from gender-based violence with level of post-traumatic stress disorder scale (DSM-V) moderate or severe,
* b) age >18 years,
* c) they could manage to stand in the position of "lying", "sitting", and "standing" without assistance

Exclusion Criteria:

* a) they could not follow the intervention due to mental or physical health

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2021-12-30 (Estimated); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in Davidson Trauma Scale (DTS) | Baseline, 1 month , 3 months and 6 months follow up
  The DTS is a 17-item self-report measure that assesses the 17 DSM-IV symptoms of PTSD. Items are rated on 5-point frequency (0 = "not at all" to 4 = "every day") and severity scales (0 = "not at all distressing" to 4 = "extremely distressing"). Respondents are asked to identify the trauma that is most disturbing to them and to rate, in the past week, how much trouble they have had with each symptom.
  The DTS yields a frequency score (ranging from 0 to 68), severity score (ranging from 0 to 68), and total score (ranging from 0 to 136). It can be used to make a preliminary determination about whether the symptoms meet DSM criteria for PTSD. Scores can also be calculated for each of the 3 PTSD symptom clusters

SECONDARY OUTCOMES:
Change in Beck Depression Inventory (BDI) | Baseline, 1 month , 3 months and 6 months follow up
  BDI consisting of 21 items with a score range from 0 to 63, with a higher score indicating a greater degree of depression.
Change in State-Trait Anxiety Inventory (STAI) | Baseline, 1 month , 3 months and 6 months follow up
  Stai with statements scoring from 1 to 4; the whole score is from 0 to 60, with higher scores indicating a greater degree of anxiety
Change in Short Form 36 (SF36) | Baseline, 1 month , 3 months and 6 months follow up
  It measured quality of life, a generic tool whose scores range from 0 to 100; higher scores denote better quality of life. It contains 36 items grouped into eight subscales: physical functioning, physical role, bodily pain, general health, vitality, social functioning, emotional role, and mental health.
Change in Visual Analogue Scale (VAS) | Baseline, 1 month , 3 months and 6 months follow up
  VAS measures subjective characteristics that cannot be directly measured. The pain is measured from 0 to 10, with 0 representing "no pain" and 10 "unbearable pain".
Change in Pittsburgh Sleep Quality Index (PSQI) | Baseline, 1 month , 3 months and 6 months follow up
  Is an instrument used to measure the quality and patterns of sleep in the older adult. It differentiates "poor" from "good" sleep by measuring seven domains: subjective sleep, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleep medication, and daytime dysfunction over the last month.The client self rates each of these seven areas of sleep. Scoring of the answers is based on a 0 to 3 scale, whereby 3 reflects the negative extreme on the Likert Scale. A global sum of "5" or greater indicates a "poor" sleeper. Although there are several questions that request the evaluation of the client's bedmate or roommate, these are not scored, nor reflected in the attached instrument.

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Bravo Navarro, PhD, Study Director — Department Nursing and Physiotherapy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bravo C, Skjaerven LH, Espart A, Guitard Sein-Echaluce L, Catalan-Matamoros D. Basic Body Awareness Therapy in patients suffering from fibromyalgia: A randomized clinical trial. Physiother Theory Pract. 2019 Oct;35(10):919-929. doi: 10.1080/09593985.2018.1467520. Epub 2018 May 3. PMID 29723080
- [Result] Madsen TS, Carlsson J, Nordbrandt M, Jensen JA. Refugee experiences of individual basic body awareness therapy and the level of transference into daily life. An interview study. J Bodyw Mov Ther. 2016 Apr;20(2):243-51. doi: 10.1016/j.jbmt.2015.10.007. Epub 2015 Oct 26. PMID 27210839